CLINICAL TRIAL: NCT00450359
Title: A Prospective Evaluation of Computer Aided Detection (CAD) in the NHS Breast Screening Programme [CADET II]
Brief Title: Computer-Aided Breast Cancer Detection in Women Undergoing Screening Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aberdeen Royal Infirmary (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Screening
Other Study IDs: ABROIN-06-MRE01-14; CDR0000534404 (Registry Identifier: PDQ (Physician Data Query)); CRUK-CADET-II; ABROIN-CADET-II; EU-20709
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2008-10

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: breast imaging study
Procedure: comparison of screening methods
Procedure: radiomammography

SUMMARY:
RATIONALE: A computer-aided detection program may help doctors find breast cancer sooner, when it may be easier to treat, in women undergoing screening mammography.

PURPOSE: This randomized clinical trial is studying how well computer-aided breast cancer detection works in women undergoing screening mammography.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare, prospectively, the breast cancer detection rate and recall rate of single reading using computer-aided detection vs standard double reading in women undergoing screening mammography.

OUTLINE: This is a prospective, randomized, multicenter study. Participants are randomized to 1 of 3 screening arms.

* Arm I (double reading): Screening mammograms are independently reviewed by two readers (i.e., radiologist or radiographer), each of whom reports on any abnormalities and decides whether a participant is recalled for further assessment or returned home to routine screening. In the event there is disagreement between the readers' findings, a third reader acts as an arbitrator by rendering an interpretation of the mammogram and making the final decision to recall the participant or return to routine screening.
* Arm II (single reading with computer-aided detection [CAD]): Screening mammograms are reviewed initially by a single reader who reports on any abnormalities. The reader then re-examines the mammogram with the aid of CAD, a system that uses computer prompts to recall suspicious features or abnormalities that may have been overlooked or previously dismissed as being normal. Based on these evaluations, a recommendation is made by the reader to either recall the participant for further assessment or return home to routine screening. If there is a discrepancy between the reader's interpretation and the CAD findings, another reader may be consulted to review the mammogram.
* Arm III (double reading followed by single reading with CAD): Screening mammograms are reviewed by double reading as in arm I followed by single reading with CAD as in arm II.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 30,000 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Currently undergoing 2-view mammography for routine breast cancer screening at any of the following participating National Health Services Breast Cancer Screening Program centers:

  * Manchester
  * Coventry
  * Nottingham
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30000 (Estimated)
Dates: Start 2006-09; Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Breast cancer detection rate
Recall rate

SECONDARY OUTCOMES:
Film reader performance using computer-aided detection

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Gilbert, MD, Study Chair — Aberdeen Royal Infirmary
Locations (4):
- United Kingdom (4):
  - Walsgrave Hospital, Coventry, England
  - Withington Hospital, Manchester, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland

REFERENCES:
- [Result] James JJ, Gilbert FJ, Wallis MG, Gillan MG, Astley SM, Boggis CR, Agbaje OF, Brentnall AR, Duffy SW. Mammographic features of breast cancers at single reading with computer-aided detection and at double reading in a large multicenter prospective trial of computer-aided detection: CADET II. Radiology. 2010 Aug;256(2):379-86. doi: 10.1148/radiol.10091899. PMID 20656831
- [Result] Gilbert FJ, Astley SM, Gillan MG, Agbaje OF, Wallis MG, James J, Boggis CR, Duffy SW; CADET II Group. Single reading with computer-aided detection for screening mammography. N Engl J Med. 2008 Oct 16;359(16):1675-84. doi: 10.1056/NEJMoa0803545. Epub 2008 Oct 1. PMID 18832239